CLINICAL TRIAL: NCT03414450
Title: A Phase 1A Dose Escalation and Phase 1B Expansion Study to Evaluate the Safety and Tolerability of ETC-1907206 in Combination With Dasatinib in Advanced Haematologic Malignancies
Brief Title: Evaluation of ETC-1907206 With Dasatinib in Advanced Haematologic Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawal requested by D3
Sponsor: EDDC (Experimental Drug Development Centre), A*STAR Research Entities (Other Government)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D3-005
Record Dates: First submitted 2018-01-14; First posted 2018-01-30 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Ph+ Acute Lymphoblastic Leukemia (Ph+ALL); Ph- Acute Lymphoblastic Leukemia (Ph-ALL); Chronic Myeloid Leukemia Accelerated Phase (CML-AP, Ph+); Chronic Myeloid Leukemia Blast Crisis (CML-BC, Ph+)
Keywords: Mnk kinase inhibitor, Mnk kinase
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase | interventions — Dasatinib

STUDY DESIGN:
Intervention Model Description: In Phase 1A, an adaptive design using the ordinal Continual Reassessment Method (oCRM) will be used to determine the MTD and RD of ETC-1907206 in combination with dasatinib.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Phase 1A) (Experimental): An adaptive design using the ordinal Continual Reassessment Method (oCRM) will be used to determine the MTD and RD of ETC-1907206 in combination with dasatinib.
  Interventions: Drug: ETC-1907206; Drug: dasatinib
- Dose Expansion (Phase 1B) (Experimental): Once the MTD and/or RD has been determined in Phase 1A, an expansion cohort will be enrolled in order to characterize the safety, PK and preliminary clinical activity of ETC-1907206 in combination with dasatinib. Subjects may continue treatment in the study until disease progression, unacceptable toxicity, withdrawal of consent or it is judged not to be in the patient's interest to continue on the study.
  Interventions: Drug: ETC-1907206; Drug: dasatinib

INTERVENTIONS:
Drug: ETC-1907206 — ETC-1907206 gelatin capsules will be dosed every other day (EOD) and contain 10 mg or 50 mg of ETC-1907206.
  Other Names: ETC-206
Drug: dasatinib — dasatinib tablets at 140 mg will be dosed every day
  Other Names: Sprycel

SUMMARY:
This study evaluates the use of ETC-1907206 in combination with dasatinib in certain types of blood cancers. The first phase of the study (1A) is designed to find the highest tolerated dose of ETC-1907206, while the second phase (1B) will assess the safety and tolerability of the recommended dose of ETC-1907206. ETC-1907206 has been designed to block the activity of an enzyme of the body known as Mnk kinase, which is thought to be involved in the development of a variety of cancers.

DETAILED DESCRIPTION:
This study consists of two parts: a Phase 1A dose escalation to identify the MTD and the RD of ETC-1907206 administered in combination with dasatinib and a Phase 1B expansion at the RD.

Phase 1A: A dose escalation with an adaptive design model using ordinal continual reassessment method (oCRM) will be used to characterise the dose toxicity curve of ETC-1907206 when administered orally every other day (EOD) under fasted conditions in combination with oral once daily dasatinib (per locally approved product prescribing instructions) in order to identify the maximum tolerated dose (MTD) and recommended dose (RD) for Phase 1B.

Phase 1B: Open-label, non-randomised, to assess preliminary clinical activity and safety of ETC-1907206 administered orally EOD under fasted conditions at the RD identified in Phase 1A, in combination with dasatinib (per locally approved product prescribing instructions).

Patients will continue in the study until disease progression, the start of new anti-cancer therapy, unacceptable toxicity, death, or the completion of 12 separate 4-week treatment cycles, whichever occurs first.

As long as the Sponsor agrees to continue treatment, patients who complete 12 cycles of treatment and have no evidence of disease progression are allowed to continue on treatment past the end of treatment (EOT) visit until there is disease progression, unacceptable toxicity, the patient decides to withdraw, or it is judged not to be in the patient's interest to continue on the study.

Malignancy assessments of the underlying disease at enrolment (blood and bone marrow), Eastern Cooperative Oncology Group (ECOG) performance status, pharmacokinetic (PK) sampling for ETC-1907206 and dasatinib, sample collection for ETC-1907206 and dasatinib biomarker analysis, and safety and tolerability assessments will be performed during the study.

ELIGIBILITY:
INCLUSION CRITERIA:

Each patient (male or female) must meet all of the following criteria to be enrolled in this study:

1. Capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements.
2. Age 18 years or older (US sites) or 21 years or older (Singapore site) at Baseline.
3. Bone marrow (BM) cytogenetic analysis with at least 20 metaphase cells, confirmed advanced haematologic malignancies in any of the 4 following disease populations at Screening:

   * CML-AP, Ph+
   * CML-BC, Ph+
   * Ph+ ALL
   * Ph- ALL with relapsed and refractory disease who have exhausted all available therapy (for patients who develop T315I mutation related resistance, the definition requires failure of ponatinib treatment if drug is accessible).
4. Meets definition for one of the following study subgroups:

   CML-AP:
   * ≥ 15% and < 30% blast in peripheral blood or bone marrow, or
   * ≥ 20% basophils in peripheral blood or bone marrow or
   * ≥ 30% blasts + promyelocytes in peripheral blood or bone marrow (but < 30% blasts) or
   * < 100 x 10^9 platelets/L in peripheral blood unrelated to therapy or
   * Cytogenetic, genetic evidence of clonal evolution and
   * No extramedullary disease.

   CML-BC:
   * ≥ 30% blasts in peripheral blood or bone marrow, or
   * extramedullary disease other than hepatosplenomegaly.

   Ph+ ALL:
   * ≥ 30% blasts in blood or bone marrow and
   * no prior history of CML.

   Ph- ALL:
   * ≥ 10% blasts in bone marrow.
5. ECOG performance status of 0 to 2 at Baseline.
6. Life expectancy of at least 3 months at Baseline.
7. Adequate organ function at Baseline, including the following (noting that repeated tests at Baseline should not be performed unless there are sufficient reasons to assume the patient would meet the inclusion criteria with re testing):

   1. Total bilirubin ≤ 1.5 x upper limit of normal (ULN), unless resulting from haemolysis or documented Gilbert syndrome.
   2. Transaminases [aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 x ULN]. [< 5 x ULN if liver infiltration with tumour present]
   3. Prothrombin time (PT) < 1.5 ULN.
   4. Calculated creatinine clearance ≥ 60 mL/min (Cockcroft and Gault formula).
   5. No clinically relevant abnormalities in the urinalysis results.
   6. Haematology:

      * Haemoglobin > 10 g/dL (transfusion allowed to reach the level)
      * Neutrophils > 1,000/µL
      * Platelets > 75,000/µL.
   7. Pancreatic status:

      * Lipase ≤ 1.5 x ULN
      * Amylase ≤ 1.5 x ULN.
8. Capable of taking oral medication and following direction regarding taking study drug (either by himself/herself or by caregiver).
9. Negative serum pregnancy test at Baseline plus a negative urine pregnancy test on Day 1, Cycle 1 prior to treatment (applies to females of childbearing potential only).
10. A minimum of 2 weeks (14 days), or 5 half-lives (whichever is shorter) since last receipt of any anti-cancer therapy (except dasatinib, hydroxyurea, anagrelide or steroids), or 4 weeks from radiation or major surgery to the first administration of the study drug.
11. All non-haematological AEs of any prior anti-cancer therapy, surgery, or radiotherapy have to be resolved to NCI CTCAE Grade ≤ 1 (except alopecia) within 2 weeks prior to starting study drug.
12. Willing to submit the blood samples and bone marrow samples for PK and pharmacodynamic (PD) analyses.

CML-AP Ph+, CML-BC Ph+, Ph- ALL, and Ph+ ALL patients with relapsed and refractory disease who have exhausted all available therapy.

Subgroup-specific intolerance definition: [Intolerance to tyrosine kinase inhibitors (TKIs) or other approved treatments for CML-AP, CML-BC and Ph+ ALL; to approved treatments for Ph- ALL] defined as:

* Non-haematologic intolerance:

Patients with Grade 3 or 4 toxicity while on therapy, or with persistent Grade 2 toxicity, unresponsive to optimal management, including dose adjustments (unless a dose reduction is not considered in the best interest of the patient if response is already suboptimal) in absence of: major haematologic response (MaHR) for accelerated phase (AP), blast crisis (BC) or Ph+ ALL patients; complete remission (CR) or complete haematological response with partial haematologic recovery of peripheral blood count (CRh) for Ph- ALL.

* Haematologic intolerance:

Patients with Grade 3 or 4 toxicity [absolute neutrophil count (ANC) or platelets] while on therapy that is recurrent after dose reduction to the lowest dose recommended by drug manufacturers in the absence of: MaHR for AP, BC or Ph+ ALL patients; CR or CRh for Ph- ALL.

NOTE: For dasatinib, non-haematologic and haematologic intolerance is defined as: CTCAE Grade > 2 requiring discontinuation.

EXCLUSION CRITERIA:

Patients meeting any of the following criteria will be excluded from the study:

1. Is a male patient with sexual partner(s) of childbearing potential who is unwilling to use a highly effective method of contraception, one of which includes a condom. Sexually active male patients must use a condom during intercourse throughout the study and for 12 weeks after the end of treatment and should not father a child in this period. A condom is required to be used also by vasectomised males in order to prevent potential delivery of the study drug via seminal fluid. Female partners of male patients must be advised to also use one of the following contraception methods:

   * intrauterine device or intrauterine system;
   * prior sterilisation; or
   * total abstinence from male/female intercourse.
2. Is a female patient of childbearing potential, defined as a female physiologically capable of becoming pregnant (including a female whose career, lifestyle, or sexual orientation precludes intercourse with a male partner, and females whose partners have been sterilised by vasectomy or other means), unless they are using a highly effective method for birth control throughout the study and for 12 weeks after the end of treatment. Highly effective methods for birth control include the following:

   * Total abstinence: This is an acceptable method when this is consistent with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   * Female sterilisation: The patient has had a surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks prior to taking study drug. In case of an oophorectomy alone, the reproductive status of the patient must have been confirmed by follow-up hormone level assessment.
   * Male partner sterilisation: The patient has the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. (For female patients on the study, the vasectomised male partner should be the sole partner for that patient.) These patients must also agree to the use an intrauterine device or intrauterine system AND a barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, or cream, or vaginal suppository. Reliable contraception must be maintained throughout the study and for 12 weeks after study drug discontinuation.
   * Females considered post-menopausal and not of childbearing potential: The definition applies to females who have had 12 months of natural (spontaneous) amenorrhoea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or 6 months of spontaneous amenorrhoea with serum follicle-stimulating hormone (FSH) levels > 40 million international units per milliliter (mIU/mL) (for US only: and estradiol < 20 pg/mL) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least 6 weeks prior to starting treatment. In the case of oophorectomy alone, only when the reproductive status of the patient has been confirmed by follow-up hormone level assessment is she considered not of childbearing potential.
3. Is a pregnant or nursing (lactating) female, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/mL).
4. Has dasatinib intolerance (haematologic and non-haematologic). Defined as: CTCAE Grade >2
5. Has received anti-cancer therapy within 2 weeks or 5 half-lives, whichever is shorter (except for hydroxyurea, steroids, allopurinol, febuxostat, rasburicase, and intravenous hydration), prior to starting study drug or the side effects of such therapy have not resolved to Grade ≤1 within 2 weeks prior to starting study drug.
6. Is receiving concomitant anti-cancer therapy (except for hydroxyurea, steroids, anagrelide, allopurinol, febuxostat, rasburicase, and intravenous hydration during the first week of the study drug[s] administration, or corticosteroids when appropriate).
7. Has used other investigational drugs within 2 weeks or 5 half-lives (whichever is shorter) prior to the first dose of study drug.
8. Has undergone autologous or allogenic stem cell transplantation < 60 days prior to the first dose of study drug;
9. Has any evidence of on-going graft-versus-host disease (GVHD).
10. Has evidence of another malignancy not in remission or history of such a malignancy within the last 3 years (except for treated basal or squamous cell carcinoma of the skin, or in situ cancer of the cervix).
11. Has central nervous system (CNS) metastases.
12. Has significant bleeding disorder unrelated to the disease.
13. Has a history of long QT syndrome or prolonged QT interval corrected based on Fridericia's method (QTcF) > 450 ms.
14. Has ECG evidence of complete left bundle branch block, or ventricular pacing.
15. Has abnormalities in the 12-lead ECG that in the opinion of the Investigator increase the risk of participating in the study (e.g., sinus rhythm with PR interval > 240 ms or second degree or higher atrioventricular (AV) block confirmed by a repeat ECG).
16. Has blood pressure and heart rate (HR) higher than 160/100 mmHg and 100 beats per minute (bpm), respectively, or lower than 80/50 mm Hg and 45 bpm, respectively, confirmed by a repeat assessment.
17. Is receiving treatment with drugs known to be associated with Torsade de Pointes.
18. Has ophthalmic signs or symptoms, such as flashes and colour perception changes.
19. Has evidence of electrolyte imbalance such as hypokalaemia, hypocalcaemia, and hypomagnesaemia of NCI-CTCAE Grade ≥ 2 (NCI CTCAE version 4.03).
20. Has symptomatic chronic heart failure; unstable angina pectoris, cardiac arrhythmia.
21. Has cardiac left ventricular ejection fraction (LVEF) < 40% (assessed by transthoracic echocardiography).
22. Has a history of myocardial infarction and/or thromboembolism in the past 6 months.
23. Has uncontrolled diabetes mellitus, neurologic or psychiatric condition, an ongoing systemic (including opportunistic) clinically significant infections or any other significant or unstable concurrent medical illness that in the opinion of the Investigator would preclude protocol therapy.
24. Has a known history of human immunodeficiency virus (HIV) sero positivity and/or is receiving combination anti retroviral therapy.
25. Has a history of gastric bypass surgery or with pre-existing gastrointestinal disorders that may interfere with proper absorption of the drug, as per Investigator's judgement.
26. Has history of seizure disorders or CNS leukaemia.
27. Is receiving cytochrome P450 3A4 (CYP3A4) inhibitors within 7 days prior to the first dose of ETC-1907206 or receiving CYP3A4 inducers within 14 days prior to the first dose of ETC-1907206 and dasatinib.
28. Cannot start treatment with dasatinib 140 mg daily, oral.
29. Is unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) (Phase 1A) | the initial 28 days of treatment
  The MTD is defined as the highest possible dose with a predicted probability of having DLT not exceeding the target toxicity rate. The target toxicity rate (or the target predicted probability of DLT) for this study is set at 25%.
Phase 1B Safety: Incidence of Adverse Events (AEs) during Phase 1B | up to 44 months
  Incidence and Severity of AEs
Phase 1B PK: Area under the drug concentration-time curve (AUC) from time zero to infinite time (AUC0-inf) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of AUC0-inf after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1B PK: AUC from time zero to the last measureable concentration (AUC0-t) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of AUC0-t after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1B PK: First-order rate constant for elimination of drug (kel) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of kel after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1B PK: Time to reach maximum plasma concentration (Tmax) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of Tmax after dosing on Day 1 and Day 15 (Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1B PK: Time between drug administration and first observed concentration above lower limit if quantitation in plasma (Tlag) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of Tlag after dosing on Day 1 and Day 15 (Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1B PK: Total clearance (CL) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of CL after dosing on Day 1 and Day 15 (Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1B PK: Volume of distribution (Vd) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of Vd after dosing on Day 1 and Day 15 (Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1B PK: Half-life (T1/2) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of T1/2 after dosing on Day 1 and Day 15 (Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).

SECONDARY OUTCOMES:
Phase 1A Safety: Incidence of Adverse Events (AEs) during Phase 1A | up to 24 months
  Incidence and Severity of AEs
Phase 1A PK: Area under the drug concentration-time curve (AUC) from time zero to infinite time (AUC0-inf) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of AUC0-inf after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1A PK: AUC from time zero to the last measureable concentration (AUC0-t) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of AUC0-t after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1A PK: First-order rate constant for elimination of drug (kel) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of kel after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1A PK: Time to reach maximum plasma concentration (Tmax) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of Tmax after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1A PK: Time between drug administration and first observed concentration above lower limit if quantitation in plasma (Tlag) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of Tlag after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1A PK: Total clearance (CL) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of CL after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1A PK: Volume of distribution (Vd) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of Vd after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1A PK: Half-life (T1/2) | pre-dose, at 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours (± 6 minutes), and at 24, 30, and 48 hours (± 2 hours) after dosing
  Single-dose PK measurement of T1/2 after dosing on Day 1 and Day 15 Cycle 1) and pre-dose on Day 1 of Cycle 2 and beyond (each Cycle is 28-days in length).
Phase 1B Clinical Activity: Best Overall Response (BOR) | through study completion (44 months)
  The BOR for each patient is determined by the following hierarchical orders:
  * For CML-AP Ph+, CML-BC Ph+ and Ph+ ALL: major molecular response, major cytogenetic response (complete response, partial response), major haematologic response (complete response, complete remission), minor haematologic response,cytogenetic response (minor response, minimal response, no response), progressive disease
  * For Ph- ALL: complete haematologic response, complete response with partial haematologic recovery, progressive disease
  The response rate will be summarised and two-sided 95% confidence intervals (CIs) on the response rates will be calculated. The best overall response will be listed.
Phase 1B Clinical Activity: objective response rate (ORR) | through study completion (44 months)
Phase 1B Clinical Activity: duration of objective response (DOR) | through study completion (44 months)
Phase 1B Clinical Activity: duration of major molecular response (DOMMR) | through study completion (44 months)
Phase 1B Clinical Activity: duration of complete haematologic response (DOCHR) | through study completion (44 months)
Phase 1B Clinical Activity: duration of complete remission (DOCRe) | through study completion (44 months)
Phase 1B Clinical Activity: duration of complete cytogenetic response (DOCCyR) | through study completion (44 months)
Phase 1B Clinical Activity: time to objective response (TTR) | through study completion (44 months)
Phase 1B Clinical Activity: time to major molecular response (TTMMR) | through study completion (44 months)
Phase 1B Clinical Activity: time to complete haematologic response (TTCHR) | through study completion (44 months)
Phase 1B Clinical Activity: time to complete remission (TTCRe) | through study completion (44 months)
Phase 1B Clinical Activity: time to complete cytogenetic response (TTCCyR) | through study completion (44 months)
Phase 1B Clinical Activity: progression-free survival (PFS) | through study completion (44 months)
Phase 1B Clinical Activity: overall survival (OS) | through study completion (44 months)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Leong, MD, PhD, Study Chair — D3 (Drug Discovery and Development)
Locations (6):
- United States (5):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided